CLINICAL TRIAL: NCT04288661
Title: The Drain Debate: Reevaluating Prophylactic Drains in Total Gastrectomy- A Controlled Trial on the Use of Prophylactic Drains in Total Gastrectomy for Gastric Cancer
Brief Title: Perianastomotic Drain After Gastrectomy (DRAG)
Acronym: DRAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: THEODOROU DIMITRIOS (Other)
Responsible Party: Sponsor-Investigator, THEODOROU DIMITRIOS, PROFESSOR, University of Athens
Organization: University of Athens (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1678 / 31-01-2020
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer
Keywords: prophylactic drain; total gastrectomy; gastric cancer; esophagogastric anastomosis leak; drain criteria
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (No Intervention): The patients of this arm undergo perianastomotic drain placement, as per standard of care institutional practice
- No drain (Experimental): The patients of this arm do not undergo perianastomotic drain placement.
  Interventions: Procedure: No drain placement

INTERVENTIONS:
Procedure: No drain placement — The need of perianastomotic drain placement after Roux-en-Y reconstruction in total gastrectomy operations is investigated. As intervention, no drain placement is considered, according to the criteria stated above
  Arms: No drain

SUMMARY:
Gastric cancer ranks as the fifth most common and fifth most lethal cancer globally. For patients with AJCC stages IB to IIIC, representing the majority of cases, the current gold standard of surgical treatment involves total gastrectomy combined with D2 lymph node dissection, followed by gastrointestinal tract reconstruction .It has long been established that minimizing surgical intervention correlates with faster patient recovery. The Enhanced Recovery After Surgery (ERAS) guidelines provide globally recognized perioperative recommendations for a variety of surgical procedures, grounded in research, audits, and evidence-based practice. In 2014, Mortensen et al. introduced ERAS guidelines specifically tailored for gastrectomy in gastric cancer. These guidelines include both procedure-specific and general recommendations applicable to the perioperative management of abdominal surgeries.Since the publication of ERAS guidelines, evidence suggests limited and inconsistent global adherence to the protocol for gastrectomy, particularly regarding surgical drain use.Drains remain in use for gastrectomy, particularly in the East, where ongoing studies explore the prognostic value of drain contents post-gastrectomy without reaching consensus. Western adherence to ERAS recommendations on drains is similarly low.This prospective, non-randomized controlled clinical trial aims to assess the impact of one perianastomotic drain when it is placed under specific, predefined criteria. The trial evaluates the immediate and short-term postoperative outcomes in patients who underwent D2 total gastrectomy for gastric cancer which were performed in a high-volume centre and under the care of a highly experienced team

DETAILED DESCRIPTION:
The DRAG (DRains After Gastrectomy) Trial is a prospective, non-randomized, controlled clinical trial involving patients diagnosed with gastric neoplasm. All surgeries were performed by a single, highly experienced surgeon in the 1st Propaedeutic Surgery Department at Hippocration General Hospital in Athens, Greece. The patients underwent open total gastrectomy with D2 lymph node dissection, followed by Roux-en-Y gastrointestinal tract reconstruction, in accordance with a predefined, ERAS-compliant perioperative departmental protocol. Our institution's protocol does not routinely incorporate exploratory laparoscopy or peritoneal cytology.

The participants were divided into two groups. The first group followed the department's standard practice, with a drain placed near the esophagojejunal anastomosis (drain group). In contrast, the second did not have a drain placed (non-drain group). The decision to place a drain was based on the following criteria:

1. Pulmonary diseases under oxygen therapy
2. Chronic oral steroid use (≥5mg/day prednisone equivalent for >1month)
3. Intraoperative hemodynamic instability requiring vasopressors
4. Intraoperative blood loss exceeding 250 mL
5. Vessel injury (celiac axis or its branches)
6. Injury to adjacent structures (pancreas, spleen, duodenum)
7. Tension of the anastomosis
8. Uncertainty regarding duodenal stump integrity due to either staple misfire or tissue quality issues Per our departmental protocol, patients were gradually mobilized starting directly after surgery, when feasible. On the second postoperative day, an oral gastrografin study was conducted for each patient to detect any early anastomotic leaks. Following a normal radiological study, patients were initiated on a liquid diet, which was then advanced to pureed food on the third postoperative day, and a soft diet on the fourth day. For patients in the drain group, the drain was removed on the fifth postoperative day, provided that the drainage volume was less than 50 mL over the preceding 48 hours, in line with departmental protocol The primary outcomes measured in this study were: a) pain levels, assessed using the Visual Analog Scale (VAS) during the first 5 postoperative days, b) postoperative nausea and vomiting (PONV) within the first 5 days, c) initiation of feeding, d) postoperative bowel mobilization, e) patient mobilization, f) length of hospital stay (LOS) Secondary outcomes included: a) mortality, b) surgically related readmissions and c) reoperations This study was conducted in accordance with the principles outlined in the Helsinki Declaration of Human Rights and with the Guidelines of Good Clinical Practice . The final study protocol and the informed consent form for participant inclusion received approval from the Institutional Review Board (IRB). The IRB also conducted regular assessments, as required, to ensure the ongoing compliance with lawful medical practice throughout the trial.

The statistical analysis was performed using the R software (R foundation for Statistical Computing) version 4.3.0 for Windows. Descriptive characteristics for the quantitative data were expressed as median and Quartile 1 (Q1) to Quartile 3 (Q3) range and for completeness reasons the mean ± standard deviation (SD), for the qualitative data was reported the frequency of occurrence and the relevant percentage. Comparisons were preformed between patients with drainage and those without drainage; for the qualitative parameters statistical tests were performed via the chi-square test (and if required a Fisher exact test) and for the arithmetic data (as normality was not possible to be ensured using the Shapiro Wilk test), were applied not parametric tests, specifically the Mann Whitney U test. The significance level (p-value) was set to 0.05, thus statistically significant difference between compared groups was for p<0.05 and all tests were two sided.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Histologically proven EGJ (Siewert II or III) or non-EGJ gastric adenocarcinoma (intestinal, diffuse, or mixed Lauren type)
* Surgical candidates for total gastrectomy plus D2 lymph node dissection
* ECOG performance status 0 or 1
* Signed informed consent from
* Preoperative evaluation of cTanyNanyM0 according to the American Joint Committee on Cancer Staging Manual, 7th edition

Exclusion Criteria:

* M1 disease
* Other unplanned organ excision
* Massive ascites or cachexia
* Current participation in any other clinical trial
* Severe cardiovascular, respiratory tract, kidney, liver, or psychiatric disease.
* Poor compliance to the clinical protocol
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Theodorou, Professor, Study Chair — University of Athens; Maria-Malvina Eleftheriou, MD, Principal Investigator — Hippocration General Hospital of Athens
Locations (1):
- Hippocration General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drain | No Drain
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drain | No Drain | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [63 to 87] | 73 [48 to 77.5] | 73 [48 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 23 | 9 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 20 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: a) Number of Participants With High Pain Levels (Using the Visual Analog Scale)
Description: Postoperative pain levels will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). VAS scores will be recorded during the patient's hospital stay following total gastrectomy. For analysis, pain intensity will be categorized into two groups:
  High pain: VAS score greater than 5
  Not high pain: VAS score 5 or less
  This binary classification will be used to compare postoperative pain outcomes between patients with and without anastomotic drain placement, helping to evaluate whether drain usage is associated with increased postoperative pain.
Time Frame: Hospital stay, an average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 31 | 3

2. Primary Outcome: Number of Participant Who Exhibited Postoperative Nausea and Vomiting (PONV) Within the First 5 Days
Description: Postoperative nausea and vomiting (PONV) is considered an immediate effect of the perianastomotic drain. Measured as present or absent, with presence meaning worse results
Time Frame: Hospital stay, an average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 24 | 5

3. Primary Outcome: Number of Participants With Delay of Feeding Initiation
Description: immediate outcome of perianastomic drain placement. Feeding is considered delayed if started after the 3rd day as per our protocol
Time Frame: Hospital stay, an average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 15 | 2

4. Primary Outcome: Number of Participants With Delay of Postoperative Mobilization
Description: immediate postoperative effect of drain placement. Mobilization is considered delayed if the patient does not manage to achieve the milestones as per our(and ERAS)protocol.
Time Frame: Hospital stay, an average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 20 | 2

5. Primary Outcome: Length of Hospital Stay
Description: immediate effect of drain placement
Time Frame: Hospital stay, an average of 5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
days | 7 [6 to 10] | 5 [5 to 6]

6. Primary Outcome: Day of Postoperative Bowel Mobilization
Description: immediate effect of drain placement. If there is no mobilization of bowel (flatus or motion) within the first 3 days, it is considered delay of the bowel movement
Time Frame: Hospital stay approx 5 days
Measure: Median (Full Range); unit: days
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
days | 4 [3 to 4] | 3 [2 to 4]

7. Secondary Outcome: Mortality
Description: short term effect of drain placement
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 1 | 2

8. Secondary Outcome: Surgically Related Readmissions
Description: short term effect of drain placement
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 5 | 0

9. Secondary Outcome: Reoperations
Description: short term effect of drain placement
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drain | No Drain
Number analyzed (Participants) | 40 | 20
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 30 days
Description: 1 adverse event:intraoperative pancreatic injury
Arm/Group | Drain | No Drain
All-Cause Mortality (participants affected / at risk) | 1/40 | 2/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/20
Other Adverse Events (participants affected / at risk) | 4/40 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drain (N=40) | No Drain (N=20)
pancreatic inlury (Surgical and medical procedures) | 0 (0) | 1 (1) — pancreatic injury/leak due to compression during lymph node dissection, detected 2 days later
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drain (N=40) | No Drain (N=20)
anastomotic leak (Surgical and medical procedures) | 4 (4) | 2 (2) — anastomotic leak
postoperative bleeding (Surgical and medical procedures) | 3 (3) | 0 (0) — Postoperative bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04288661/Prot_SAP_000.pdf